CLINICAL TRIAL: NCT03361787
Title: Efficacy of a Multi-dimensional Program for Parents of Adolescents With High-functioning Autism
Brief Title: A Multi-dimensional Program for Parents of Adolescents With High-functioning Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0269-17-HMO-CTIL
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder
Keywords: adolescents; parents; coaching
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parentship coaching intervention (Experimental)
  Interventions: Behavioral: "Parentship"- a multi dimensional intervention program to improve parental resilience

INTERVENTIONS:
Behavioral: "Parentship"- a multi dimensional intervention program to improve parental resilience — "Parentship" is a multi dimensional intervention program to improve parental resilience and adolescent participation using the OPC model.

SUMMARY:
The purpose of this pilot study is to examine the initial efficacy of a multi-dimensional coaching intervention ("Parentship") for parents of adolescents with High Functioning Autism (HFASD).

The "Parentship" protocol is a short-term intervention program in occupational therapy that aims to promote parental resilience and enhance adolescents' participation in daily life.

DETAILED DESCRIPTION:
"Parentship" is a structured occupational therapy intervention for promoting parental resilience and enhance adolescents' participation in daily life The Parentship protocol uses OPC (Graham & Rodger, 2010) as the primary treatment approach. Its primary goal is to lead parents into recognition and understanding of their adolescent's multi-dimensional personal profile that includes sensorimotor, cognitive-behavioral, and social-communicative and personal factors, as required by the International Classification of Functioning (ICF) model (WHO, 2007).

The intervention will be administered by occupational therapists on an individual (or both parents) basis, once a week, over 3-4 months.

10-15 families will be recruited through community advertising. Data will be collected at the onset and completion of the intervention. Data will be analysed using quantitative and qualitative methods.

Adverse events, if occur, will be reported to supervising neurologist and the Helsinki Committee.

ELIGIBILITY:
Inclusion Criteria:

* ASD diagnosed by certified medical practitioner
* parent report regarding barriers to occupational performance/participation
* SP2 or BRIEF-Parent or SSIS scores reflecting at least 1 SD from typical

Exclusion Criteria:

* Diagnoses of severe neurological or psychiatric health condition.
* Instability in pharmacological treatment

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 3-4 months
  structured interview administered by occupational therapist
Autism: Parenting Questionnaire (APQ) | 3-4 months
  7 dimensions (Knowledge About Autism, Communication, Play, Behaviour Management, Confidence, Stress Management, and Family Functioning) are the focus of this questionnaire that serves as a basis for intervention with parents

SECONDARY OUTCOMES:
Clinical Assessment of Therapeutic Responses (CATR) | 1.5 months and 3 months
  a questionnaire that monitors the abilities of the therapist to create an optimal parent-therapist relationship

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical organization, Jerusalem Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided